CLINICAL TRIAL: NCT04563637
Title: A Comparison of Computer Vision Based Approach vs. Dual Energy X-ray Absorptiometry Scan to Measure Body Fat
Brief Title: A Comparison of Computer Vision Based Approach vs. Dual Energy X-ray Absorptiometry Scan to Measure Body Fat Percentage
Status: Terminated | Type: Observational
Why Stopped: Sponsor terminated due to lack of funding
Sponsor: Centennial Medical Group (Industry)
Responsible Party: Sponsor
Other Study IDs: U1111-1250-0418
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Computer Based Vision: A 15 second long video will be obtained at the research site using a smart phone or tablet. Then subjects will undergo a whole body dual energy x-ray absorptiometry scan . Then the subject will go home and take a second 15 second long video. The videos will then be analyzed by computer based vision application and the body fat percentage measured by dual energy x-ray absorptiometry scan will be compared.
  Interventions: Diagnostic Test: Computer based vision application by video; Radiation: whole body dual energy x-ray absorptiometry scan

INTERVENTIONS:
Diagnostic Test: Computer based vision application by video — patients will be tested by computer based analysis of a video as well as by dexa scan.
Radiation: whole body dual energy x-ray absorptiometry scan — subjects will receive a whole body dual energy x-ray absorptiometry scan to measure their body fat percentage
  Other Names: Dexa scan

SUMMARY:
This study is being done to test whether a HealthReel computer vision-based software application can estimate body fat percentage with equivalent accuracy to a whole body dual energy x-ray absorptiometry scan.

DETAILED DESCRIPTION:
This study is being done to test whether a computer vision-based software application can estimate body fat percentage with equivalent accuracy to a whole body dual energy x-ray absorptiometry scan. The dual energy x-ray absorptiometry scan involves lying on a machine for about 6-10 minutes. It is an open design. The study will also examine whether waist circumference measurement improves the accuracy of the body fat percentage estimate by the computer vision-based application.A total of approximately 492 subjects are planned to take part in this study at one study center.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to provide informed consent before any trial-related activities
* Male or female, age > = 18 at time of signing informed consent
* Have access to and ability to use a smart phone to take a 15 second video from their home

Exclusion Criteria:

* Pregnancy at the time of screening
* Known osteoporosis with a T-score of <-2.5 at hip or spine or pathological fracture of spine
* Cirrhosis of the liver, or presence of ascites

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males and Females are eligible to participate, based on their biologic identity.
Study Population: Males and females between ages 18 and 100
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
variance in body fat percentage between computervision application and dexa scan | 8 months
  Variance between body fat percentage measured by smart phone applicaiton compared to body fat percentage as measured by DEXA scan

SECONDARY OUTCOMES:
abdominal circumference | 8 months
  Analysis will be undertaken to see if the variance between application and dual energy x-ray absorptiometry is reduced when the abdominal circumference is included in the application or whether inclusion of abdominal circumference does not reduce the variance.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Geller, Principal Investigator — Centennial Medical Group
Locations (1):
- Centennial Medical Group, Elkridge, Maryland, United States

IPD SHARING:
Plan to Share IPD: No